CLINICAL TRIAL: NCT02662751
Title: The Impact of Performing a Low-dose, Whole-body Angiography as the First Element of an Imaging Assessment Following Stroke or Transient Ischemic Attack in Comparison With Usual Care: a Randomized, Controlled, Open Trial
Brief Title: Performing a Low-dose, Whole-body Angiography as the First Element of an Imaging Assessment Following Stroke / TIA
Acronym: VASCU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AOI/2014/FM-01; 2015-A01600-49 (Other: RCB number)
Record Dates: First submitted 2015-11-17; First posted 2016-01-26 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Ischemic Attack, Transient
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Imaging (Active Comparator): Patients randomized to this arm will have routine post-stroke/TIA imaging assessments.
  Intervention: Routine Imaging Assessment
  Interventions: Other: Routine Imaging Assessment
- LDWBA first (Experimental): Patients randomized to this arm will start their post-stroke/TIA imaging assessment by a low-dose, whole-body angiography (LDWBA). The latter can be followed by routine imaging assessments if required.
  Intervention: LDWBA first followed by Routine Imaging Assessment if required.
  Interventions: Other: Routine Imaging Assessment; Device: LDWBA first (CT scan)

INTERVENTIONS:
Other: Routine Imaging Assessment — Patients will have the usual post-stroke/TIA imaging assessment according to routine procedures in each participating center. The latter most often begin with an angiography of the supra-aortic trunks but may also include a range of other imaging exams depending on the patient's condition.
  "Routine Imaging Assessment" refers to an imaging strategy and not a specific device. The devices used depend on what is available in participating centres and the routine choices made by those centers.
Device: LDWBA first (CT scan) — Patients randomized to this arm will start their post-stroke/TIA imaging assessment by a low-dose, whole-body angiography (LDWBA). The latter can be followed by routine imaging assessments if required.
  LDWBA: This is a low dose scanner protocol comprising a CT acquisition and an iodine contrast medium injection. The acquisition includes a propeller during the arterial phase of the contrast agent injection in the cervical and thoracic levels with cardiac gaiting (ECG gating to reduce cardiac motion artifacts), continuing with pelvic abdominal arterial acquisition. The second propeller is made on the abdomen and pelvis at the portal time of injection. The reconstruction will be carried out in pulmonary, mediastinal and bone windows. The dose will be calculated for each patient.
  Arms: LDWBA first

SUMMARY:
The main objective of this study is to compare two post-stroke/TIA (transient ischemic attack) imaging strategies in terms of the number of clinically important (i.e. requiring specific treatment according to current recommendations) lesions detected. The first strategy is the current/usual strategy in each participating centre and the second strategy consists in starting the post-stroke/TIA imaging assessment by a whole-body, low-dose angiography and subsequently resorting to elements of the usual strategy if required.

DETAILED DESCRIPTION:
The secondary objectives are:

A. To compare the patient pathways between the two arms in terms of time to diagnosis, and duration of hospitalization.

B. To compare the consumption of imaging exams (number and type) and total body irradiation between the two arms.

C. To compare the diagnostic efficiency between the two arms in terms of detection of predefined lesions, and performance ratios.

D. To study the thickness of the left atrial wall as a risk factor for permanent atrial fibrillation.

E. To compare the distribution of suspected neoplasms between the two groups, as well as the number of detected incidentalomas.

F. To compare the survival and the incidence of new cardiovascular events between the two arms at 12 months and 36 months.

G. To compare the quality of life between the two arms at 12 months and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* The patient was informed about the implementation of the study, its objectives, constraints and patient rights
* The patient has given free and informed consent and signed the consent
* Patient affiliated with or beneficiary of a health insurance plan
* Patient available for 36 months of follow-up
* The patient has had a stroke (within the past 10 days, diagnosis confirmed by MRI with a diffusion sequence) or transient ischemic attack (within the past 10 days, ABCD2 score greater than 3) without haemorrhage

Exclusion Criteria:

* The patient is currently participating in or has participated in another biomedical research study within the past three months or is currently in an exclusion period determined by a previous study.
* Patient under guardianship or judicial protection
* Refusal to sign the consent
* Inability to correctly inform the patient or his/her trusted person about the study
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contraindication for a treatment used in this study
* Known allergy to contrast medium or severe allergy to iodine
* Known active malignancy or history of cancer treatment
* The patient has already undergone a full body scanner in the previous three months
* Renal failure with creatinine clearance below 60 ml / min
* Monoclonal immunoglobulin
* History of severe symptomatic cardiovascular event (myocardial infarction, aortic dissection, mesenteric ischemia, renal ischemia)
* Emergency situations that hamper the planned course of the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Presence/absence of at least one element requiring specific treatment | Day 30
  This is a binary variable: the units are "presence/absence".
  Presence/absence of at least one element (found during the patient's pathway in the imaging service) requiring specific treatment from among the following:
  * Anomaly indicating a high risk for cardio-vascular embolism
  * Anomaly indicating a high risk for vascular thrombosis
  * Any other lesions requiring specific treatment

SECONDARY OUTCOMES:
Diagnostic delay (h) | between day 1 and hospital discharge (expected maximum of two weeks)
  The time lapsed between inclusion in the study and the first etiological determination of a diagnosis.
  Thus units (h) is consistent with the time frame.
Length of hospital stay (h) | hospital discharge (expected maximum of two weeks)
  The units are given in hours even for long stays.
Patient pathway: the number of imaging exams required | Month 1
Patient pathway: the types of imaging exams required | Month 1
Total irradiation (mSv) during patient pathway | Month 1
For contrast injections during the patient pathway: total grams of iodine injected | Month 1
Number of atherosclerotic sites detected / number of imaging examinations performed | Month 1
The presence / absence of tight stenosis on the supra aortic arteries | Month 1
The presence / absence of an occlusion on the supra aortic arteries | Month 1
The presence / absence of a dissection on the supra aortic arteries | Month 1
The number of atherosclerotic lesions in the aortic arch | Month 1
For each atherosclerotic lesion in the aortic arch: plaque thickness (mm) | Month 1
For each atherosclerotic lesion in the aortic arch: presence/absence of crevices | Month 1
For each atherosclerotic lesion in the aortic arch: presence/absence of plaque thromboses | Month 1
Detection of patent foramen ovale (yes/no) | Month 1
Presence / absence of a thrombus or a circulatory stasis in the left atrium | Month 1
Extent of atherosclerosis: affects the coronary arteries? yes/no | Month 1
Extent of atherosclerosis: affects the aortic valve? yes/no | Month 1
Extent of atherosclerosis: affects the aortic arch? yes/no | Month 1
Extent of atherosclerosis: affects the abdominal aorta? yes/no | Month 1
Extent of atherosclerosis: affects the renal arteries? yes/no | Month 1
Extent of atherosclerosis: affects digestive arteries? yes/no | Month 1
Extent of atherosclerosis: affects iliac or common femoral arteries? yes/no | Month 1
Extent of atherosclerosis: affects supra aortic trunks? yes/no | Month 1
For each detected incidentaloma: volume (mm^3) | Month 1
The thickness of the left atrial wall | Month 1
Presence / absence of paroxysmal atrial fibrillation | 36 months
Presence / absence of a cardiovascular event de novo. | 36 months
  Presence / absence of a cardiovascular event de novo. The following events will be searched for:
  * New stroke or TIA
  * Major Cardiovascular Events (acute symptomatic vascular disease)
Survival (yes/no) | 12 months
Survival (yes/no) | 36 months
EQ-5D-5L questionnaire | 12 months
EQ-5D-5L questionnaire | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Macri, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes